CLINICAL TRIAL: NCT00367731
Title: Neurological Outcomes With in THAI National HAART Program.
Brief Title: NOW Thai HAART Study
Status: Completed | Type: Observational
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Rajavithi Biomolecular Research Center (Other)
Other Study IDs: RVH_CER_003
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2006-08-23 (Estimated); Status verified 2006-08

CONDITIONS: HIV; AIDS; Neurological Complications
Keywords: HIV; AIDS; Neurological complications; HAART
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Drug: Highly Active Antiretroviral Treatment (combination of :NRTI, NNRTI,or PI)

SUMMARY:
After Initiation of HAART in peoples who living with HIV/AIDS in Thailand by the year 2000, rapidly expanded HAART access of national project has been promoted in 2004. Free ARVs (For CD4<200cell/cu.mm. or in symptomatic HIV with CD4<250 cell/cu.mm. )and CD4 monitoring has been available. The first-line regimen is d4T+3TC+NVP in mainly the first time (Naive) patients. CD4 response ), rate of opportunistic infection, and neurological outcomes were measured. Rate of ARV change, adverse events,treatment failure, TB co-infection rate, percent changing to EFV-based regimen or PI-based regimen were recorded.

Any Adverse Events including, Sever rash, Severe Hepatitis, Lipid abnormalities, Severe Anemia and Other, common AEs will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* HIV/AIDS patients.
* Age >15 years.
* informed consent

Exclusion Criteria:

* Not informed consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 2005-01; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Subsai Kongsaengdao, M.D., Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (3):
- Thailand (3):
  - Rajavithi Hospital, Bangkok
  - Lumpang Hospital, Lumpang
  - Sappasithiprasong Hospital, Ubonratchathani